CLINICAL TRIAL: NCT01946841
Title: Effets de la Nutrition entérale spécifique RealDiet®Renal (NES) Chez Des Patients Insuffisants rénaux hémodialysés dénutris : efficacité, tolérance, qualité de Vie.
Brief Title: Specific Enteral Nutrition in Malnourished, Dialysis Patients With Chronic Kidney Disease. Efficacy, Safety, Quality of Life
Acronym: AL-EN-PHED
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Patient recruitment
Sponsor: Lactalis (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRD - 2013 - ALENPHED
Record Dates: First submitted 2013-08-06; First posted 2013-09-20 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Kidney Disease; Renal Failure Chronic Requiring Hemodialysis; Severe Malnutrition; Tolerance; Quality of Life; Activity; Appetite and General Nutritional Disorders
Keywords: Chronic kidney disease; Hemodialysis; Severe malnutrition; Enteral nutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Malnutrition; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RealDiet®Renal enteral nutrition (Experimental)
  Interventions: Dietary Supplement: RealDiet®Renal

INTERVENTIONS:
Dietary Supplement: RealDiet®Renal

SUMMARY:
The objective of this unblinded study is to assess the nutritional effects of a 12 weeks administration of the specific enteral nutrition (SEN) RealDiet®Renal pockets, as well as the impact on the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patient on hemodialysis for at least 3 months, with a minimum of three hemodialysis sessions of 4 hours per week
* Patients aged 18 years
* Written, free and informed consent given by the Patient
* Patient insured under the social security system or equivalent
* Patients who did not receive enteral nutrition during the 3 months preceding inclusion ; taking an oral nutritional supplement, or per-dialytic parenteral nutrition or total parenteral nutrition is not a criterion of non-inclusion
* Patient in a state of malnutrition

  * defined by the presence of at least 3 out of 5 of the following criteria :

    * weight loss greater than 10% observed in the last six months
    * serum albumin <35 g / l
    * serum Prealbumin <300 mg / l
    * BMI <20
    * NPNA <1 g / kg / day for 2 consecutive months

and

* presenting

  * food intake <20 kcal / kg / day or
  * failure of other nutritional care methods, namely, oral nutritional supplements and / or peridialytic parenteral nutrition, or total parenteral nutrition
  * lack of compliance after one month, to the nutritional care methods mentioned above. • Patients for whom the decision to prescribe enteral feeding was previously taken

Exclusion Criteria:

* Patients with a history of intolerance to enteral feeding
* Index Kt/Veq (balanced) < or = 1.2 or index Kt/Vsp (single pool) < or = 1.4 according to the method used
* Patients with a disease compromising the short-term (4-6 months) prognosis (cancer or other disease in the terminal phase)
* Pregnant Patient
* Patient with a known allergy to at least one of the following : milk protein, soy, fish
* Patient whose digestive tract is not functional or patient in shock
* Patient protected under guardianship
* Patient in exclusion period after participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evolution of serum prealbumin and albumin. | 6 months
  Evaluate during 3 months specific enteral nutrition (SEN) treatment, and 3 months after treatment interruption, the effects of the study product on the evolution of serum prealbumin and albumin.

SECONDARY OUTCOMES:
Evolution of nutritional status during 3 months of enteral nutrition, and during 3 months after end of treatment. | 6 months
Evolution of quality of life during 3 months of enteral nutrition, and during 3 months after end of treatment. | 6 months
Evolution of tolerance of study product during 3 months of enteral nutrition. | 3 mois

CONTACTS AND LOCATIONS:
Locations (1):
- Lactalis, Retiers, France